CLINICAL TRIAL: NCT00774462
Title: FORCE: Rituximab (CD 20+-B Cell-depleting Monoclonal Antibody) for the Treatment of Refractory Inflammatory Myopathies With Specific Antibodies and Refractory Myasthenia Gravis
Brief Title: Rituximab for the Treatment of Refractory Inflammatory Myopathies and Refractory Myasthenia Gravis
Acronym: FORCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P051204
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2007-12

CONDITIONS: Myositis; Myasthenia Gravis
Keywords: Myositis; Anti-synthetase; Anti-SRP; Myasthenia gravis; Rituximab
MeSH Terms: conditions — Myositis; Myasthenia Gravis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab 1000 mg intravenous, 2 times, 2 weeks apart and 1000 mg 6 months after the last injection

SUMMARY:
The traditional treatment of inflammatory myopathies (IM) and generalized myasthenia gravis (MG) is immunosuppressive therapy, usually beginning with corticosteroids. However, up to 70% of treated patients show an incomplete response, including 10 - 30% who are unresponsive. Corticosteroids and other immunosuppressive therapies presented also many side effects. We propose to evaluate in a pilot, open, prospective, multicentric, phase II study, the interest of rituximab in the treatment of patients with primary IM associated with specific AAb (anti-synthetase and anti-SRP AAbs), or MG (with anti-AchR AAbs), refractory to conventional therapies. Twenty fourth patients with primary IM (12 with anti-synthetase, 12 with anti-SRP AAbs), and 12 with MG will be included in the study.

DETAILED DESCRIPTION:
Rituximab, a chimeric monoclonal antibody specific for human CD20, which targets B lymphocytes, has been first developed as biotherapy for the treatment of B lymphoma. In this context, hundred thousands patients received this drug, with a very good tolerance. Recently, interest has grown in the pivotal role of B cells for auto-immune humorally mediated diseases. Rituximab could then be a potential new biological treatment for such diseases, especially for patients refractory to conventional therapies. As a Muscular Diseases Centre, we have a large recruitment of patients with inflammatory myopathies (IM) and myasthenia gravis (MG). Although the physiopathogenesis of these two conditions differ, both can be associated with specific auto-antibodies (AAbs) and their therapeutic management is almost similar. The traditional treatment approach to IM and generalized MG is immunosuppressive therapy, usually beginning with corticosteroids. However, up to 70% of treated patients show an incomplete response, including 10 - 30% who are unresponsive. We propose to evaluate in a pilot, open, prospective, multicentric, phase II study, the interest of rituximab in the treatment of patients with primary IM associated with specific AAb (anti-synthetase and anti-SRP AAbs), or MG (with anti-AchR AAbs), refractory to conventional therapies.

Inclusions criteria are IM (as defined by the 119th European Neuromuscular Centre workshop) or generalised MG (as defined by the Texas Clinical Classification System) associated with specific AAbs (anti-synthetases (JO1, PL7 or PL12), or anti-SRP for primary IM, and anti-AchR for MG) and refractory to conventional treatments defined as an inadequate response to, or intolerable side effects with conventional treatments, such as corticosteroids, azathioprine, methotrexate, cyclophosphamide, cyclosporine, IgIV and/or plasma exchange.

The therapeutical schema is rituximab 1000 mg, 2 times (at day 0 and 15), followed by one single injection (1000 mg) 6 months latter and end of follow up at 1 year.

The efficacy is evaluated by an improvement of Kendall's muscular testing or MG muscular score at month 12. Secondary criteria include Kendall's muscular testing or MG muscular score at day 21 and month 7, quality of life auto-questionnaire (SF 36), evolution of CK levels and AAb titers.

Twenty fourth patients with primary IM (12 with anti-synthetase, 12 with anti-SRP AAbs), and 12 with MG will be included in the study. If a success is observed in at least 6 patients, it will be possible to conclude that the response rate is above 25% (lower 90% confidence interval for observed response rate 50%).

ELIGIBILITY:
Inclusion Criteria:

* For myositis III. Idiopathic myositis

  1. Myositis as defined by the 119th ENMC:

     1. Proximal myopathy with weakness
     2. Subacute or insidious onset over 18 years
     3. Myogenic syndrome on EMG (optional)
     4. Muscle fibre necrosis and regeneration and/or inflammatory cell infiltrate on muscular biopsy
  2. Specific AAbs : anti-synthetases (anti-JO1, anti-PL7, or anti-PL12), or anti-SRP.

     IV. Refractory to the conventional treatments Resistance to conventional treatments is defined as an inadequate response to, or intolerable side effects with conventional treatments, such as corticosteroids, azathioprine, methotrexate, cyclophosphamide, cyclosporine, IgIV and/or plasma exchange. At least one or more of these drugs or therapeutical approaches (used alone or as a combination) must have been unsuccessfully tested before inclusion. Inadequate response is defined as the lack of improvement and/or the degradation of evaluation parameters (defined bellow) despite these conventional therapies, that led to a modification or a reintroduction of treatment.
* For myasthenia III. Generalised MG

Generalised seropositive MG as defined by the Texas Clinical Classification System:

1. Extraocular muscle weakness quantified with MG muscle score (MMS), whose inter and inter observer reproducibility has been demonstrated [44].
2. Specific AAbs : anti-AchR IV. Refractory to the conventional treatments Resistance to conventional treatments is defined as an inadequate response to, or intolerable side effects with conventional treatments, such as corticosteroids, azathioprine, methotrexate, cyclophosphamide, cyclosporine, IgIV and/or plasma exchange. At least one or more of these drugs or therapeutical approaches (used alone or as a combination) must have been unsuccessfully tested before inclusion. Inadequate response is defined as the lack of improvement and/or the degradation of evaluation parameters (defined bellow) despite these conventional therapies, that led to a modification or a reintroduction of treatment

Exclusion Criteria:

* Other muscular diseases, such as:

  1. Inclusion body myositis
  2. Macrophagic myofasciitis
  3. Inherited myopathies
* Secondary IM to one other connective tissue disorders

  1. Systemic scleroderma (ARA and/or "LEROY AND MEDSGER" criteria)
  2. Sjögren's syndrome (European criteria)
  3. Systemic lupus erythematosus (ACR criteria)
  4. Rheumatoid arthritis (ACR criteria)
  5. Mixed connective tissue disease (ACR criteria)
* Other myasthenic syndrome, such as:

  1. Non generalised, ocular MG
  2. Lambert Eaton syndrome
  3. MG associated with malignant thymoma
  4. Inherited myasthenic syndrome
* Cancer (or cancer-associated myositis)
* Age < 18 years
* Pregnancy
* HIV seropositivity
* Evolutive infection (B, C hepatitis, tuberculosis)
* Lack of approved consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Score of muscular strength (Kendall's muscular testing for myositis or MG muscular score for myasthenia) | at month 12

SECONDARY OUTCOMES:
- Score of muscular strength (Kendall's muscular testing for myositis or MG muscular score for myasthenia) | at day 21 and month 12
- Improvement of functional scale score (SF36) | at day 21 and month 12
- Decrease of CK levels | at day 21 and month 12
- Evolution of auto-antibody titers | at day 21 and month 12
- Improvement of extra-muscular activity of the disease such as the level of lung involvement by pulmonary function tests | at day 21 and month 12
- Improvement in the treatment burden defined as the possibility to decrease the dose or stop some of the drugs used at entry | at day 21 and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BENVENISTE, PUPH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service de Médecine Interne 1 / Groupe Hospitalier Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Derived] Allenbach Y, Guiguet M, Rigolet A, Marie I, Hachulla E, Drouot L, Jouen F, Jacquot S, Mariampillai K, Musset L, Grenier P, Devilliers H, Hij A, Boyer O, Herson S, Benveniste O. Efficacy of Rituximab in Refractory Inflammatory Myopathies Associated with Anti- Synthetase Auto-Antibodies: An Open-Label, Phase II Trial. PLoS One. 2015 Nov 5;10(11):e0133702. doi: 10.1371/journal.pone.0133702. eCollection 2015. PMID 26539981